CLINICAL TRIAL: NCT04023708
Title: A Pregnancy Registry to Evaluate the Safety of Dengue Vaccine Among Inadvertently Exposed Pregnant Women and Their Offsprings (DNG16)
Brief Title: Observational Study to Evaluate the Safety of CYD Tetravalent Dengue Vaccine (CYD-TDV) in Pregnant Women and Their Offsprings Inadvertently Exposed During Pregnancy
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DNG16; U1111-1217-3443 (Registry Identifier: ICTRP)
Record Dates: First submitted 2019-06-27; First posted 2019-07-17 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Dengue Virus Infection
MeSH Terms: conditions — Dengue | interventions — Dengue Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Biospecimen Retention: None Retained — No biospecimens will be collected from participants, therefore, no biospecimens will be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort I: CYD-TDV exposed pregnant women and offspring: Pregnant women of any age and their offspring who were inadvertently exposed to CYD-TDV anytime during the pregnancy or in the 30 days preceding their LMP
  Interventions: Drug: CYD-TDV Dengue Vaccine

INTERVENTIONS:
Drug: CYD-TDV Dengue Vaccine — Pharmaceutical form:Solution Route of administration: Intramuscular
  Other Names: Dengvaxia®

SUMMARY:
Primary Objective:

To evaluate the safety of CYD-TDV in pregnant women and their offsprings inadvertently exposed during pregnancy or up to 30 days preceding their last menstrual period (LMP) with regards to maternal, pregnancy, birth, neonatal and infant outcomes. Specifically, the frequency/rates of these outcomes will be: (i) described, and (ii) compared with population-level background incidence rates prior to the introduction of CYD-TDV immunization (i.e., external unvaccinated comparator).

Secondary Objective:

To describe:

* the characteristics of women exposed to CYD-TDV during pregnancy or up to 30 days before the LMP
* the characteristics of CYD-TDV pregnancy exposure with regards to number of doses, dose intervals, and trimester of exposure.

DETAILED DESCRIPTION:
This is a non -interventional (observational) post authorization safety study (PASS): no vaccine will be administered as part of the study.

This pregnancy registry study is a combination of a retrospective (outcomes occurred before the start of participant enrollment) and prospective (outcomes occurred after the start of participant enrollment) cohort study using active identification and enrollment of pregnant women and their offsprings inadvertently exposed to CYD-TDV during pregnancy or up to 30 days preceding the LMP.

The study period will be from July 2016 (first availability of Paraná's Immunization Registry) to July 2022 (end of last follow-up interview for offsprings), and the participant enrollment period will last approximately 1 year.

Study duration per participant will vary depending on: 1) the stage of pregnancy at the time the participant will be enrolled; 2) whether the participant will be included retrospectively or prospectively. The maximum duration will be 22.5 months (up to 9 months of pregnancy + 42 days post-delivery [puerperium period] + 12 months post-birth).

ELIGIBILITY:
Inclusion criteria:

* CYD-TDV exposed pregnant women of any age residing in the 30 municipalities of Paraná where public vaccination campaigns have been offered at the time of their pregnancy exposure, and whose pregnancy exposure was reported to Brazil's AEFI PV database (SI-PNI AEPV).
* Valid contact information (in SI-PNI AEPV).
* Study participants must provide a signed and dated informed consent form (ICF) or assent form (AF) (based on local regulations), and/or a signed and dated ICF by the parent(s) or other legally acceptable representative (and by an independent witness if required by local regulations) if a minor (women who meet the inclusion criteria and provide informed consent to participate and complete the structured interview, but who do not consent to medical record review and/or database linkages will still be included in the study; however, their data will be analyzed separately in a sensitivity analysis).

Exclusion criteria:

- Presence of a major language barrier, medical or psychiatric condition that would prevent a woman from providing informed consent or accurate medical or medication/vaccination histories.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible pregnant women of any age residing in Paraná who received at least one dose of CYD-TDV during pregnancy or up to 30 days preceding LMP and the offsprings resulting from those pregnancies. The study could also be extended to other regions and states of Brazil.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Percentage of pregnant women with maternal adverse events | From cohort entry up to 42 days post-end of pregnancy
  Maternal adverse events defined as all reported adverse events following immunization (serious and non-serious) occurring independent of the pregnancy (e.g., injection site reactions, systemic reactions)
Percentage of pregnant women with pregnancy related adverse events | From cohort entry to up to 42 days post-end of pregnancy
  Pregnancy related adverse events defined as adverse event of special interest (AESI)s and other reported adverse events (serious and non-serious) occurring during the pregnancy, labour and delivery, or the puerperium
Percentage of offsprings with adverse birth outcomes | On day of birth (DOB)
  Adverse birth coutcomes defined as study AESIs and other reported adverse events (serious and non-serious) observed or diagnosed at birth
Percentage of offsprings with adverse neonatal events | From DOB up to 28 days post-birth
  Adverse neonatal events defined as study AESIs and other reported adverse events (serious and non-serious) occurring between DOB and 28 days post-DOB
Percentage of offsprings with adverse infant events | From day 29 post-birth up to 12 months post-birth
  Adverse infants events defined as study AESIs and other reported adverse events (serious and non-serious) occurring between day 29 post-birth and 12 months post-birth

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Universidade Federal do Paraná Site Number : 1, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://www.vivli.org/